CLINICAL TRIAL: NCT02671929
Title: Translation and Development of an Online Self-help Intervention With Subsequent Feasibility Study as an After Care After Inpatient Psychosomatic Treatment
Brief Title: Translation and Development of an Online Self-help Intervention With Subsequent Feasibility Study
Acronym: KEN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Dr. Rüdiger Zwerenz, Principle Investigator, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RK-91809
Record Dates: First submitted 2016-01-15; First posted 2016-02-02 (Estimated); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Treatment Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- self-help program + feedback (Experimental): Patients in this arm receive access to the internet-based self-help program and get feedback on their progress in the program.
  Interventions: Behavioral: self-help program; Behavioral: therapeutic feedback
- self-help program (Active Comparator): Patients in this arm receive access to the internet-based self-help program and don't get any therapeutic feedback
  Interventions: Behavioral: self-help program

INTERVENTIONS:
Behavioral: self-help program — Access to the internet-based self-help program
Behavioral: therapeutic feedback — Therapeutic feedback on the written information sent to the online therapist
  Arms: self-help program + feedback

SUMMARY:
The purpose of this study is to determine the feasibility and effectiveness of an internet-based self help program concerning satisfaction with the treatment and their life, depression and anxiety. Both study groups get access to the internet-based self-help program. The intervention group receives additional feedback to their progress in the program from an online therapist. The investigators hypothesize that (1) at least 75% of the patients in the intervention group are "satisfied" or "very satisfied" with the self-help program, (2) 50% of the patients in the intervention group work with all eight units and (3) patients of the intervention group have a higher emotional competence than the patients of the control group at the end of the self-help program.

ELIGIBILITY:
Inclusion Criteria:

* day care/ inpatient treatment in the Department of Psychosomatic Medicine and Psychotherapy at the University Medical Center of the Johannes Gutenberg-University Mainz
* minimum age of 18 years
* private internet access
* e-mail address

Exclusion Criteria:

* acute suicidality
* psychosis
* current alcohol or drug addiction
* life time diagnosis of a schizophrenic, schizoaffective, bipolar or organic psychic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-09; Primary Completion 2016-05 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Satisfaction of the intervention group with the internet-based self-help program measured with an reworded version of the "patient satisfaction questionnaire" (ZUF-8) | 10 weeks after study inclusion (T1)

SECONDARY OUTCOMES:
Emotional competence measured with the "SEK-27" (questionnaire for self-assessment of emotional competence) | 10 weeks after study inclusion (T1) and 19 weeks after study inclusion (T2)
Depression measured with the German version of the "PHQ-9" (Patient Health Questionnaire) | 10 weeks after study inclusion (T1) and 19 weeks after study inclusion (T2)
Quality of life measured with the German version of the "EUROHIS-QOL 8" (European Health Interview Survey Quality of Life 8) | 10 weeks after study inclusion (T1) and 19 weeks after study inclusion (T2)
Anxiety measured with the German version of the "GAD-7" (General Anxiety Disorder Screener) | 10 weeks after study inclusion (T1) and 19 weeks after study inclusion (T2)
Self-esteem measured with the German version of the "RSE" (Rosenberg Self-Esteem Scale) | 10 weeks after study inclusion (T1) and 19 weeks after study inclusion (T2)
Somatoform afflictions measured with the German version of the "SSS-8" (Somatic Symptom Scale) | 10 weeks after study inclusion (T1) and 19 weeks after study inclusion (T2)
Subjective prognosis of work ability measured with the "SPE" (Subjective Prognosis of Work Ability) | 10 weeks after study inclusion (T1) and 19 weeks after study inclusion (T2)
Therapeutic alliance measured with the German version of the "WAI-SR" (Working Alliance Inventory - Short Revised) | 10 weeks after study inclusion (T1)
Depersonalisation measured with the German short version of the "CDS-2" (Cambridge Depersonalisation Scale) | 10 weeks after study inclusion (T1) and 19 weeks after study inclusion (T2)
Acceptance of the internet-based self-help program measured with an especially for the self-help program devised questionnaire | End of every unit (weekly) and 10 weeks after study inclusion (T1)
Usage of the internet-based self-help program measured with an especially for the self-help program devised questionnaire | 10 weeks after study inclusion (T1)
Utilization of alternative after care measures (psychotherapy and drugs) with a self-devised questionnaire | 10 weeks after study inclusion (T1)

CONTACTS AND LOCATIONS:
Overall Officials: Manfred E Beutel, Prof. Dr., Study Director — Department for Psychosomatic Medicine and Psychotherapy at the University Medical Center of the Johannes Gutenberg-University Mainz
Locations (1):
- University Medical Center, Department of Psychosomatic Medicine and Psychotherapy, Johannes Gutenberg University, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zwerenz R, Becker J, Johansson R, Frederick RJ, Andersson G, Beutel ME. Transdiagnostic, Psychodynamic Web-Based Self-Help Intervention Following Inpatient Psychotherapy: Results of a Feasibility Study and Randomized Controlled Trial. JMIR Ment Health. 2017 Oct 16;4(4):e41. doi: 10.2196/mental.7889. PMID 29038094